CLINICAL TRIAL: NCT02384642
Title: Creating Opportunities Through Mentoring, Parenting and Safe Spaces - a Randomized Controlled Trial in Democratic Republic of Congo
Brief Title: Creating Opportunities Through Mentoring, Parenting and Safe Spaces - Democratic Republic of Congo
Acronym: COMPASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: International Rescue Committee (Other); Department for International Development, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Lindsay Stark, Associate Professor of Population and Family Health, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAO6612
Record Dates: First submitted 2015-02-24; First posted 2015-03-10 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Sexual Assault; Interpersonal Relations; Marital Status; Domestic Violence
Keywords: Adolescent Health; Democratic Republic of Congo; Sexual Violence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- COMPASS (Active Comparator): The COMPASS program will involve a structured intervention for girls between the ages of 10-14 that is intended to engage adolescent girls, those who are influential in their lives, service providers and other stakeholders, with the ultimate goal of co-creating environments in which girls are valued and safe. The program is centered on establishing or supporting community-supported safe spaces for girls where they can come and gather among themselves and participate in a structured life-skills curriculum.
  Interventions: Behavioral: COMPASS
- COMPASS plus parenting (Experimental): In the COMPASS plus parenting intervention arm, girls will receive the COMPASS intervention, and In addition to the safe spaces for girls, the COMPASS project will also implement structured activities for the parents and caregivers of participants. The study will examine the relative impact of the parenting initiative in addition to the program for adolescent girls. The study will seek to determine whether the structured intervention with girls' parents has an added impact on outcomes improve girls' safety and well-being.
  Interventions: Behavioral: COMPASS plus parenting

INTERVENTIONS:
Behavioral: COMPASS — COMPASS (Creating Opportunities through Mentoring, Parental involvement and Safe Spaces) is a program for 10-14 year old girls in Eastern DRC. The program is a structured intervention that is intended to engage adolescent girls, through life skills training and establishing or supporting community-supported safe spaces for girls where they can come and gather among themselves and participate in a structured life-skills curriculum.
  Arms: COMPASS
Behavioral: COMPASS plus parenting — The COMPASS plus parenting intervention is the core COMPASS intervention, plus activities for the parents and caregivers of participants.
  Arms: COMPASS plus parenting

SUMMARY:
The study is a randomized controlled trial of COMPASS, an intervention for adolescent girls in Eastern Democratic Republic of Congo. The study design will employ a two-arm randomized controlled trial where girls will be enrolled at the same time and randomized to receive a basic package of services, which includes life skills education and access to mentors in safe spaces, or the basic package plus a structured parenting intervention for girls' caregivers. An experimental design will be used to evaluate the relative impact of the parenting initiative in addition to the safe space program for girls. In addition, qualitative research will address additional questions of acceptability, processes of change and best practice.

Groups in North and South Kivu will be randomized so that every group is randomly designated as a group that will either roll out the core intervention or the intervention plus caregiver component. Groups that do not receive the parental intervention during the study will receive the intervention when the study is complete to reduce communal jealousies.

The intervention, the COMPASS program, will involve a structured intervention for girls between the ages of 10-14 that is intended to engage adolescent girls, those who are influential in their lives, service providers and other stakeholders, with the ultimate goal of co-creating environments in which girls are valued and safe. The program is centered on establishing or supporting community-supported safe spaces for girls where they can come and gather among themselves and participate in a structured life-skills curriculum. In addition to the safe spaces for girls, the COMPASS project will also implement structured activities for the parents and caregivers of participants.

DETAILED DESCRIPTION:
The study will examine the relative impact of the parenting initiative in addition to the program for adolescent girls. The study will seek to determine whether the structured intervention with girls' parents has an added impact on outcomes improve girls' safety and well-being. Research will focus on unpacking the components of the program in order to determine which components or combination of components have the most impact. This research will include a mix of qualitative and quantitative approaches to establish a foundation for good programming that supports adolescent girls' safe and healthy transition into adulthood.

The study assessment will employ a mixed methods approach with most data collection occurring at pre-test/baseline and post-intervention, although a qualitative assessment will also be performed at the intervention midpoint as a process indicator. Quantitative survey methods will be used to evaluate attitudes towards a host of topics related to physical and financial assets and health-related behaviors. Survey questions will be administered using Audio Computer Assisted Self-Interviewing (ACASI) and Computer-Assisted Personal Interviewing (CAPI). Quantitative methods will be used to yield statistical measures of the scale of changes in attitudes, skills, and behaviors due to the intervention.

Qualitative methods will include in-depth semi-structured interviews and focus group discussions with girls, their family members and mentors, as well as participatory methods with girls to assess topics such as self-esteem, empowerment, and resilience.

ELIGIBILITY:
Inclusion Criteria:

* female
* aged 10-14
* give informed consent

Exclusion Criteria:

- cognitive impairment

Ages: 10 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1633 (Actual)
Dates: Start 2015-06; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Sexual violence in the past 12 months | 12 months
  A binary composite representing any form of sexual violence in the previous 12 months, which included self-reported forced sex, unwanted sexual touching, or coerced sex

SECONDARY OUTCOMES:
Change in baseline prevalence of interpersonal relationships | 12 months
  This study will use a questionnaire to measure whether there is an increase in study participants' average number close friends from the pre-test to post-test evaluation. Girls will also self-report sources of emotional support such as comfort in discussing problems with a trusted female adult and comfort discussing topics such as education, marriage, puberty, pregnancy prevention, HIV/AIDS, and financial plans with caregivers
Change in baseline prevalence of physical abuse | 12 months
  This study will use a questionnaire to measure whether the percentage of girls who self-reported experiencing beatings within the past 12 months decreases between the pre-test and post-test evaluation
Change in baseline prevalence of early marriage | 12 months
  This study will use a questionnaire to measure changes in the percentage of girls who self-reported being married from the pre-test to post-test evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Stark, Principal Investigator — Associate Professor of Population and Family Health
Locations (1):
- International Rescue Commitee, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Seff I, Falb K, Yu G, Landis D, Stark L. Gender-equitable caregiver attitudes and education and safety of adolescent girls in South Kivu, DRC: A secondary analysis from a randomized controlled trial. PLoS Med. 2021 Sep 28;18(9):e1003619. doi: 10.1371/journal.pmed.1003619. eCollection 2021 Sep. PMID 34582454
- [Derived] Stark L, Seff I, Asghar K, Roth D, Bakamore T, MacRae M, Fanton D'Andon C, Falb KL. Building caregivers' emotional, parental and social support skills to prevent violence against adolescent girls: findings from a cluster randomised controlled trial in Democratic Republic of Congo. BMJ Glob Health. 2018 Oct 19;3(5):e000824. doi: 10.1136/bmjgh-2018-000824. eCollection 2018. PMID 30398222
- [Derived] Stark L, Seff I, Assezenew A, Eoomkham J, Falb K, Ssewamala FM. Effects of a Social Empowerment Intervention on Economic Vulnerability for Adolescent Refugee Girls in Ethiopia. J Adolesc Health. 2018 Jan;62(1S):S15-S20. doi: 10.1016/j.jadohealth.2017.06.014. PMID 29273113
- [Derived] Falb KL, Tanner S, Ward L, Erksine D, Noble E, Assazenew A, Bakomere T, Graybill E, Lowry C, Mallinga P, Neiman A, Poulton C, Robinette K, Sommer M, Stark L. Creating opportunities through mentorship, parental involvement, and safe spaces (COMPASS) program: multi-country study protocol to protect girls from violence in humanitarian settings. BMC Public Health. 2016 Mar 5;16:231. doi: 10.1186/s12889-016-2894-3. PMID 26945586